CLINICAL TRIAL: NCT00982475
Title: Ablation at St. George Hospital - Prospective Randomized Comparison of Manual and Mechanical Remote Robotic Catheter Ablation for Drug-Refractory Atrial Fibrillation
Brief Title: Alster Man and Machine: Comparison of Manual and Mechanical Remote Robotic Catheter Ablation for Drug-Refractory Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Kai Jaquet (Industry)
Collaborators: Abbott Medical Devices (Industry); Hansen Medical (Industry)
Responsible Party: Sponsor-Investigator, Dr. Kai Jaquet, Prof. Dr. Roland Richard Tilz, Asklepios proresearch
Organization: Asklepios proresearch (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1889
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Atrial Fibrillation
Keywords: pulmonary vein isolation; robotic navigation; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PVI with robotic navigation (Active Comparator)
  Interventions: Procedure: Pulmonary vein isolation with radiofrequency current
- PVI manually (Placebo Comparator)
  Interventions: Procedure: Pulmonary vein isolation with radiofrequency current

INTERVENTIONS:
Procedure: Pulmonary vein isolation with radiofrequency current — Pulmonary vein isolation with radiofrequency current

SUMMARY:
Long term results after pulmonary vein isolation (PVI) with robotic navigation in patients with drug refractory atrial fibrillation are not inferior to manual radiofrequency current ablation.

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal atrial fibrillation
* persistent atrial fibrillation < 2 month
* indication for catheter ablation
* LEF > 50%
* diameter LA < 50 mm

Exclusion Criteria:

* intracardial thrombus
* atrial fibrillation with underlying curable disease
* renal failure > stage I
* contraindication for anticoagulation
* life expectancy < 12 month
* previous PVI
* pregnancy

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-09; Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Freedom of AF 12 months after procedure. | 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- ASKLEPIOS KLINIK St. Georg, Hamburg, Germany

REFERENCES:
- [Derived] Rillig A, Schmidt B, Di Biase L, Lin T, Scholz L, Heeger CH, Metzner A, Steven D, Wohlmuth P, Willems S, Trivedi C, Galllinghouse JG, Natale A, Ouyang F, Kuck KH, Tilz RR. Manual Versus Robotic Catheter Ablation for the Treatment of Atrial Fibrillation: The Man and Machine Trial. JACC Clin Electrophysiol. 2017 Aug;3(8):875-883. doi: 10.1016/j.jacep.2017.01.024. Epub 2017 Jun 28. PMID 29759785